CLINICAL TRIAL: NCT05386134
Title: Adaptive Optics Imaging in Retinal Disorders
Brief Title: Adaptive Optics Retinal Imaging in Inherited and Acquired Retinal Disorders
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Ajoy Vincent, Associate Professor, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000078905
Record Dates: First submitted 2022-04-14; First posted 2022-05-23 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Genetic Disease; Inherited Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Subjects: Approximately 175 Study Subjects
  Interventions: Device: Adaptive Optics Retinal Camera
- Control Group: Approximately 25 Control group
  Interventions: Device: Adaptive Optics Retinal Camera

INTERVENTIONS:
Device: Adaptive Optics Retinal Camera — The rtx1 is a non-invasive device functions without making contact with the eye. The fundus of the patient's eye is illuminated with the IR light emitted from the illumination optical system. The device is comprised of an optoelectronic sensor (OES) that measures the optical defects, software that calculates the necessary corrections and a deformable mirror (DM) that constantly adapts its shape to restore the image's clarity. The digital camera, which is built into the instrument, receives the images and then the images are recorded in the computer hard disk. The AO image software registers and averages the captured image series in order to reduce noise and produce a final enhanced image. The rtx1 integrates AO technology in a flood illumination imaging system and enables visualizing the retina with a high transverse optical resolution of 250 line-pairs per millimeter.

SUMMARY:
This is a Prospective Observational study. The aim of the study is to understand the underlying photoreceptor, retinal pigment epithelium or retinal vascular aberrations in inherited and acquired retinal disorders. The study would use adaptive optics (AO) technology to assist in-vivo visualization of these retinal structures and ascertain changes from normal. Further, by using the AO imaging in patients before and after treatments, this study aims to better understand the effect of various interventions and develop AO as an outcome measure in various retinal disorders.

DETAILED DESCRIPTION:
The investigators plan to recruit approximately 200 participants (approximately 175 study subjects and 25 Control group) having an inherited or acquired retinal disease. The study participants will be screened based on Inclusion and exclusion criteria. Eligible study and control participants will be consented prior to conducting any study related procedures. For the Data Collection, patient information including previous eye examination, past medical history and family history will be obtained from hospital charts. Patients will be asked to return for a follow-up visit at 6-months and at 1 year.

The Objectives of the study include:

1. To test AO imaging in patients with well characterized genetic and non-genetic diseases in an attempt to - To better understand the underlying photoreceptor, retinal pigment epithelium or retinal vascular aberrations - To utilize the AO imaging in patients before and after treatments to better understand the effect of the intervention and develop AO as an outcome measure in various retinal disorders
2. To test AO in healthy controls to serve as internal controls Patients with inherited or acquired retinal disease who satisfy the inclusion criteria and those who consent for the study will be screened for the study. Study participants and participants from the cohort group will then have a 6 month or annual follow-up visit as per the study protocol.

The primary outcome measures will be the quantify cone photoreceptors (density and spacing), retinal pigment epithelium density and retinal blood vascular flow in retinal disorders and compare it with controls. This will be calculated using software algorithms incorporated within AO machine (rtx1). Patient data will be compared with age-matched control data.

The secondary outcome measure would be to ascertain if using rtx1, the rate of progression of retinal disease or treatment effect can be quantified. To accomplish this, areas that were imaged at baseline will be reimaged at the follow up visits. Since the rtx1 machine has the capability to identify exact retinal location between the visits, these follow up images will be compared to baseline images to determine rate of disease progression or effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Aged 5 - 70 years
3. Diagnosed with well documented retinal disorder

Control group Inclusion Criteria:

1. Subjects aged 5 years - 70 years with normal eye examination.
2. Patients with strabismus and otherwise normal visual acuity and eye examination
3. Patients with unilateral eye diseases such as cataract, with a normal eye exam in the fellow eye.

Exclusion Criteria:

1. Inability of the subject to maintain a stable position while seated
2. Uncontrolled nystagmus, trembling or movements of the eyes or the head
3. Presence of cataract or any opacity in the front of the eye that obscures retinal imaging
4. Any general disease such neurological disease which could affect vision and the retina.
5. History of previous uveitis, glaucoma, previous intra-ocular surgery or photodynamic therapy
6. High refractive errors (> +15D or < -15D) that cannot be corrected by the adaptive optics system.
7. Patients who have a history of photosensitivity or take any medicine that cause photosensitivity as a side effect
8. Patients who are aphakic after cataract surgery

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Initial contact with all study participants will be by their regular ophthalmologist during a regular clinic visit. All study participants will be explained the study objectives and procedures in detail by an investigator not involved in their direct care.
  Patients with retinal dystrophies will be recruited through the Ocular Genetics Program (OGP) at the Hospital for Sick Children. Patients with acquired retinal disorders will be recruited from the pediatric retina clinic at the Hospital for Sick Children.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2032-06-13 (Estimated); Study Completion 2033-06-13 (Estimated)

PRIMARY OUTCOMES:
To measure the change in Quantification of cone receptors | Primary outcome will be measured at Baseline, 6-months ,1 year. The patient data will be compared to the control data.
  The primary outcome measures will be to measure the change in the quantification of cone photoreceptors (density and spacing).This will be calculated using software algorithms incorporated within AO machine (rtx1).
To measure the change in Quantification of the retinal pigment epithelium density | Primary outcomes will be measured at Baseline, 6-months ,1 year. The patient data will be compared to the control data.
  The primary outcome measure will be to measure the change in quantification of the retinal pigment epithelium density. This will be calculated using software algorithms incorporated within AO machine (rtx1).
To measure the change in Quantification of retinal blood vascular flow in retinal disorders | Primary outcomes will be measured at Baseline, 6-months ,1 year. The patient data will be compared to the control data.
  The primary outcome measures the wall-to-lumen ratio (WLR) and the vascular wall cross-sectional area (WSCA) of retinal arterioles.

SECONDARY OUTCOMES:
To measure the change and rate of progression of retinal disease | Secondary outcomes will be measured at follow-up visits. They will be compared to Baseline visits and measured at 6-months interval and a year
  The secondary outcome measure would be to ascertain if using rtx1, the rate of progression of retinal disease or treatment effect can be quantified. To accomplish this, areas that were imaged at baseline will be reimaged at the follow up visits. Since the rtx1 machine has the capability to identify exact retinal location between the visits, these follow up images will be compared to baseline images to determine rate of disease progression or effectiveness of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ajoy Vincent, MS, Principal Investigator — Associate Professor
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared as part of a cohort (pertaining to specific genetic disorders). This will include age, sex, genetic variant, retinal photographs and adaptive optics images.
Supporting Information: Study Protocol
Time Frame: 2026 onwards two years after the end of the study. All published literature will be accessible to researchers from the time of publication.
Access Criteria: All Researchers
URL: https://clinicaltrials.gov/study/NCT05386134?term=adaptive%20optics&checkSpell=&rank=6